CLINICAL TRIAL: NCT05644119
Title: Periodontal and Orthodontic Outcomes of Straight Versus Looped Fixed Retainers: a Split-mouth Randomized Controlled Trial
Brief Title: Periodontal and Orthodontic Outcomes of Straight vs. Looped Fixed Retainers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Talal Zahid, Associate Professor | Chairman, Department of Periodontics, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 084-09-22
Record Dates: First submitted 2022-11-19; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Orthodontic Appliance Complication; Orthodontic Appliance Design; Orthodontic Treatment
Keywords: Orthodontic retention; Fixed orthodontic retention; Fixed orthodontic retainer; V- loop bonded retainer

STUDY DESIGN:
Intervention Model Description: Split-mouth Design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- V-looped Wire Retainer (LWR) (Experimental): The LWR is a 0.569-mm (0.022-inch) Blue Elgiloy (soft) round wire (RMO). The retainer will extend from the left canine to the right central incisor.
  Interventions: Device: V- loop Bonded Orthodontic Retainer
- Straight Wire Retainer (SWR) (Active Comparator): The SWR is 0.8-mm twisted stainless steel wire (3M Unitek, Monrovia, Calif). The retainer will extend from the right canine to the left central incisor.
  Interventions: Device: Straight Wire Retainer

INTERVENTIONS:
Device: V- loop Bonded Orthodontic Retainer — The V- loop bonded retainer is a unique design that not just provides tooth stability but also allows flossing with ease.
  Other Names: V-loop Bonded Lingual Retainer; Wave Orthodontic Retainer
  Arms: V-looped Wire Retainer (LWR)
Device: Straight Wire Retainer — The straight wire retainer is a fixed bonded orthodontic retainer. This involves attaching a metal wire to the back of the teeth to keep it in position.
  Arms: Straight Wire Retainer (SWR)

SUMMARY:
The goal of this split-mouth, head-to-head, randomized controlled trial is to compare the effects of a fixed straight retainer with the V- loop bonded retainer on periodontal health in patients with the requirement of continuous fixed retention for 12-24 months after orthodontic treatment.

The main question it aims to answer is whether the V- loop bonded retainer is more effective than fixed straight retainer for periodontal health management.

Each patient will receive 2 lower fixed and bonded retainers: (1) a straight wire retainer (SWR) and (2) a looped wire retainer (LWR). Patients will be asked to floss once daily with a thread flosser.

Researchers will compare the effects of two types of retainers to see if there is a statistically significant difference.

DETAILED DESCRIPTION:
Ensuring alignment stability is a major challenge for orthodontists following an orthodontic treatment. This has led to the development of various orthodontic retention methods to enhance stability. Both fixed and removable retainers have been in use for years. However, most orthodontists nowadays prefer fixed bonded retainers over removable ones due to their many advantages, including easy to wear, being patient compliance free, long-term usability and stability, and better aesthetics. Over the past decades, many variations of fixed retainers have been developed. Of these, the current gold standard is the straight type flexible spiral (multistranded) wire retainer. Nevertheless, a major concern of using fixed straight retainers is the potential for periodontal health compromise. They are known to make oral hygiene maintenance more difficult for the patient, which in turn may lead to periodontal diseases due to more plaque and calculus accumulation. The wave or V- loop bonded retainer may be a solution to this problem, as it provides stability of teeth yet allows flossing with ease.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of continuous fixed retention for 12-24 months after orthodontic treatment
* Good periodontal health (i.e., no clinical attachment loss and < 10% bleeding on probing)

Exclusion Criteria:

* History of oral prophylaxis in the past 6 months
* History of any systemic illness such as diabetes
* Preexisting or post-orthodontic periodontal disease
* Current intake of antibiotic and/or anti-inflammatory medications
* Smoking
* Pregnancy

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of retainer failures and teeth stability through clinical examination | Approximately 2 years
  The examination will be carried out for each participant to assess the final outcome of bonds of assigned intervention immediately following the orthodontic treatment and after intervals of six months and two years.
Measurement of the Little's Irregularity Index to assess the crowding of Mandibular anterior arch | Approximately 2 years
  The examination will be carried out for each participant to assess the final outcome assigned interventions immediately following the orthodontic treatment and after intervals of six months and two years.
  The scale of the index includes the following:
  * 0: Perfect Alignment
  * 1-3: Minimal Irregularity
  * 4-6: Moderate Irregularity
  * 7-9: Severe Irregularity
  * 10: Very Severe Irregularity
  The value represents the total horizontal displacement of the anatomical contact points of the mandibular anterior teeth in millimeters.

SECONDARY OUTCOMES:
Change from Baseline (immediately following the orthodontic treatment) in gingivitis on the 4-point Modified Gingival Index (MGI) at the short-term (6 months) and long-term (2 years) | Approximately 2 years
  The MGI is a non-invasive visual instrument designed to evaluate the progression of gingivitis. The scale ranges from 0 (normal gingiva) to 3. (severe inflammation with tendency to spontaneous bleeding). Change = (Year 2 Score - Baseline Score)
Change from Baseline (immediately following the orthodontic treatment) in plaque accumulation on O'leary Plaque Index (PI) at the short-term (6 months) and long-term (2 years) | Approximately 2 years
  The PI is a valid and reliable assessment tool that records the presence of mineralized deposits and soft debris on all 4 surfaces of every tooth. It utilizes a rating scale from 0 (no plaque) to 1 (plaque present at gingival margin). Change = (Year 2 Score - Baseline Score)
Change from Baseline (immediately following the orthodontic treatment) in gingival bleeding on the Gingival Bleeding Index (GBI) by Ainamo and Bay at the short-term (6 months) and long-term (2 years) | Approximately 2 years
  The GBI is a reliable measure of periodontal stability. It uses delicate probing of the gingival sulcus orifice. Using a standardized periodontal probe with a 0.6 mm tip and 1 mm marking, the bleeding on probing (BOP) will be evaluated. A skilled examiner will measure BOP using probes with 0.25 N or less of force (25 g). If bleeding starts within 10 seconds, a positive finding is recorded.
Change from Baseline (immediately following the orthodontic treatment) in oral hygiene questionnaire at the short-term (6 months) and long-term (2 years) | Approximately 2 years
  Participants will be adminstered a self-reported oral hygiene questionnaire on brushing and flossing frequency, patient satisfaction with the retainers, and ease of flossing to determine their overall satisfaction with the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Talal Zahid, M.S, Principal Investigator — Associate Professor, King Abdulaziz University
Locations (1):
- King Abdulaziz University, Department of Periodontics, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No